CLINICAL TRIAL: NCT05765136
Title: The Effects of the Close Collaboration With Parents Training and Single-family Room Architecture on the Length of Stay and Growth Parameters of Preterm Infants - a National Multicenter Study in Finland
Brief Title: Care Outcomes in Preterm Infants Following the Implementation of Family-centered Interventions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Professor Liisa Lehtonen, Principal Investigator, University of Turku
Other Study IDs: VVM_LOS_2021
Record Dates: First submitted 2021-09-01; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: Prematurity
Keywords: Infant, preterm; Length of stay; Neonatal intensive care; Postnatal growth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Close collaboration group: Preterm infants born in hospitals where the Close Collaboration with Parents training program has been successfully implemented
- Single-family room group: Preterm infants born in hospitals that have implemented an architectural change to single-family room design
- Control group: Preterm infants born in hospitals that have not gone through any of the two aforementioned interventions (single-family room architecture or Close Collaboration with Parents training program)

SUMMARY:
The proposed study evaluates the effects of two family-centered interventions on the length of stay and outpatient visits and growth of preterm infants.The interventions are 1) the Close Collaboration with Parents training for the staff and 2) moving from traditional neonatal intensive care unit architecture to single-family room architecture.

DETAILED DESCRIPTION:
The Close Collaboration with Parents training targeted to the health care team of neonatal intensive care units to facilitate parental involvement in infant care and to support parenting. The training program involves a structured education process, where trained mentors educate staff in neonatal units. The duration of the training program is 18 months per unit. The training program has been implemented in eleven neonatal units in Finland since 2009; another 12 units haver not gone through the training.

The other intervention, single-family room architecture, provides facilities for parents to stay in the room of their infant throughout there 24 hour day. This intervention has been carried out in four neonatal units in Finland since 2014; in one by restructuring the existing unit, and in three by building a new unit/hospital.

In this study, the investigators are going to use national, population-based registers (the Medical Birth Register, the small Preterm Infant Register and the Hospital Discharge Register) governed by the Finnish National Institute for Health and Welfare. These registers have been widely used for observational studies, and contain data on all newborn infants in the country.

There are currently 23 neonatal units in Finland. Three units have undergone both interventions, nine units have undergone one intervention, and 12 units have undergone neither. Preterm infants (born before 35 gestational weeks) discharged from any unit will be divided into those who have been cared for all, part or no time in a hospital with an intervention, separately for each intervention. The outcome measures of interest will be related to health care utilization such as the length of stay and unscheduled outpatient visits, and to clinical outcomes such as postnatal growth parameters.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants (gestational age <35 weeks) born in Finland between 2006 and 2020

Exclusion Criteria:

* Missing data on key variables (gestational age, place of birth, length of stay)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Complete preterm birth cohort included in the national Medical Birth Register
Sampling Method: Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Length of stay | Immediately after discharge
  The length in days on the initial hospitalization following preterm birth

SECONDARY OUTCOMES:
Weight | Immediately after discharge
  Kilograms
Length | Immediately after discharge
  Centimeters
Head circumference | Immediately after discharge
  Centimeters
Postnatal emergency visits | Within the first year of life (corrected gestational age) after discharge home
  Amount of unplanned emergency outpatient visits after discharge from initial hospitalization
Postnatal emergency hospitalizations | Within the first year of life (corrected gestational age) after discharge home
  Duration of unplanned emergency outpatient hospitalizations after discharge from initial hospitalization
Gestational age at discharge | Immediately after discharge
  The corrected gestational age of the infant at final discharge from neonatal care

CONTACTS AND LOCATIONS:
Overall Officials: Liisa Lehtonen, Professor, Principal Investigator — Turku University Hospital and University of Turku
Locations (1):
- University of Turku, Turku, Finland

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/36/NCT05765136/Prot_SAP_000.pdf